CLINICAL TRIAL: NCT05682742
Title: A Prospective, Multicenter Clinical Investigation of the da Vinci Surgical System
Brief Title: Clinical Investigation of the da Vinci Surgical System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1097341C
Record Dates: First submitted 2022-12-22; First posted 2023-01-12 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Thymoma; Mediastinal Tumor; Gynecologic Disease; Gynecologic Cancer; Pelvic Organ Prolapse; Prostate Disease; Prostate Cancer; Inguinal Hernia; Ventral Hernia; Obesity, Morbid
MeSH Terms: conditions — Thymoma; Mediastinal Neoplasms; Genital Diseases, Female; Pelvic Organ Prolapse; Prostatic Diseases; Prostatic Neoplasms; Hernia, Inguinal; Hernia, Ventral; Obesity, Morbid | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Robotic-assisted surgery (Experimental): Subjects scheduled to undergo robotic-assisted surgery
  Interventions: Device: Robotic-assisted Surgery

INTERVENTIONS:
Device: Robotic-assisted Surgery — Subjects scheduled to undergo robotic-assisted surgery

SUMMARY:
This prospective, multicenter, single-arm study is being conducted to confirm safety, effectiveness, and usability of da Vinci Surgical System in performing robotic-assisted surgical procedures.

ELIGIBILITY:
Pre-operative Inclusion Criteria:

* Age 21 years or older
* Per study Investigator's discretion, subject is a suitable candidate to undergo multiport robotic-assisted surgery for the study specified procedure as a primary procedure

Pre-operative Exclusion Criteria:

* Subject is pregnant or suspected to be pregnant or breastfeeding
* Subject has any other condition or personal circumstance that, in the judgment of the Investigator, might interfere with the collection of complete quality data
* Subject is currently participating in or has participated in a study of an investigational agent or a significant risk investigational device study within the past 6 months
* Subject belongs to vulnerable population.
* Subject is contraindicated for anesthesia or surgery
* Subject has had previous neoadjuvant therapy, previous chemotherapy, immunotherapy, and/or radiation therapy for treatment of the cancer to be resected within the past 6 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of conversion | Intra-operative
  Effectiveness defined as the ability to complete the planned da Vinci robotic-assisted procedures without conversion to open.

SECONDARY OUTCOMES:
Incidence of adverse events | 30-day follow-up
  Safety defined as the incidence of all intra-operative and post-operative adverse events that occur through the 30-day follow-up period.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Orlando Health, Inc., Orlando, Florida
  - Sparrow Health System, Lansing, Michigan
  - The Valley Hospital, Ridgewood, New Jersey
  - The Ohio State University Wexner Medical Center, Columbus, Ohio

REFERENCES:
- [Derived] Merritt RE, Teixeira A, Needleman B, Meara M, Cosgrove C, Sanchez AE, Herrera LJ, Kwasny L, Miller R, Bartley J, Qandeel H, Levy J, Culligan P. A prospective, nonrandomized clinical investigation of the da Vinci surgical system model IS5000. J Robot Surg. 2025 Oct 1;19(1):650. doi: 10.1007/s11701-025-02837-w. PMID 41032176